CLINICAL TRIAL: NCT07368894
Title: Assessing the Effectiveness of Screening, Brief Intervention, and Referral to Treatment (SBIRT) With Personalized Feedback Intervention to Reduce Polysubstance Impaired Driving in Young Adults Aged 18-30
Acronym: ADAPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Brittney Hultgren, Assistant Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00023076; U01CE003725 (NIH); Project 7744 (Other Grant/Funding Number: Insurance Institute of Highway Safety)
Record Dates: First submitted 2026-01-20; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Impaired Driving

STUDY DESIGN:
Intervention Model Description: All participants will receive the brief online intervention. Half will be randomized to receive it immediately after baseline, the other half will receive it 3 months after baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist control (Active Comparator): Individuals will have received SBIRT but will be on a waitlist to receive the brief personalized intervention for 3 months after baseline assessment.
  Interventions: Behavioral: Personalize Feedback Intervention
- Active Intervention (Experimental): Participants will have received SBIRT and receive the brief online personalized intervention immediately after baseline assessment.
  Interventions: Behavioral: Personalize Feedback Intervention

INTERVENTIONS:
Behavioral: Personalize Feedback Intervention — The brief online personalized feedback intervention (PFI) is adapted from the personalized feedback provided in BASICS, iCHAMP, studies using similar standalone PFI approaches. Specifically, feedback adapted from these brief motivational interventions and prior projects include: Patterns of use: alcohol, cannabis, other drug, and polysubstance use frequency, alcohol and cannabis quantity and peak; Substance use norms; Expectancies of use of alcohol ; Estimates on money the participant spends on alcohol and cannabis compared; Protective behavioral strategies; Alcohol- and/or cannabis-impaired driving norms; Wait time to drive and related psychoeducation; Additional psychoeducation is provided (e.g., standard drink; information on tetrahydrocannabinol (THC) percentages) throughout the feedback to improve understanding and motivation for change.

SUMMARY:
The current study is assessing the effects of receiving Screening, Brief Intervention and Referral to Treatment alone versus also receiving a brief online personalized intervention on impaired driving behaviors among Washington State young adults aged 18-30.

DETAILED DESCRIPTION:
The current project is inviting young adult aged 18-30 in Washington State who screen at moderate or moderate to high risk or who report impaired driving during Screening, Brief Intervention and Referral to Treatment. Consented young adults would be randomized to receive a brief online personalized intervention or waitlist control and be assessed at enrollment and 3 months later. A selection of participants will be assessed at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30 at enrollment
* Received Screening, Brief Intervention, and Referral to Treatment (SBIRT) in the past 3 month
* Through SBIRT screened at moderate or moderate-to-high risk based on substance use OR reported any impaired driving the past 6 months
* Lives in Washington State
* Received a study information card from an SBIRT provider
* Consents to having Zip Code use for analyses
* Consents to randomization to receive brief online personalized intervention or waitlist control

Exclusion Criteria:

* Not meeting eligibility criteria
* Inability to confirm participant's identity, residency, or date received SBIRT.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of times in the past 3 months participants drove impaired by both alcohol and cannabis at 3 month follow-up | From baseline to 3 months later at 3 month follow up assessment.

SECONDARY OUTCOMES:
Number of times in the past 3 months participants drove impaired by both alcohol and cannabis at 6 month follow-up | From 3 month after completing baseline to 3 months later at the 6 month follow-up assessment
Number of times in the past 3 months participants drove impaired by alcohol only at 3 month follow-up | From baseline to 3 months later at 3 month follow-up assessment
Number of times in the past 3 months participants drove impaired by cannabis only at 3 month follow-up | From baseline to 3 months later at 3 month follow-up assessment
Number of times in the past 3 months participants drove impaired by alcohol only at 6 month follow-up | From 3 months after baseline to 3 months later at 6 month follow-up assessment
Number of times in the past 3 months participants drove impaired by cannabis only at 6 month follow-up | From 3 months after baseline to 3 months later at 6 month follow-up assessment
Reported wait time to drive after using both alcohol and cannabis measured in minutes at 3 month follow up | From baseline to 3 months later at 3 month follow up assessment.
  Question asks: How long do you typically wait to drive after using alcohol and Cannabis used at the same time so that the effects overlap. Participants answer in hours and minutes which is transformed into total number of minutes.
Reported wait time to drive after using alcohol measured in minutes at 3 month follow up | From baseline to 3 months later at 3 month follow up assessment.
  Question asks: How long do you typically wait to drive after using alcohol. Participants answer in hours and minutes which is transformed into total number of minutes.
Reported wait time to drive after using cannabis measured in minutes at 3 month follow up | From baseline to 3 months later at 3 month follow up assessment.
  Question asks: How long do you typically wait to drive after using cannabis. Participants answer in hours and minutes which is transformed into total number of minutes.
Reported wait time to drive after using both alcohol and cannabis measured in minutes at 6 month follow up | From 3 months after baseline to 3 months later at 6 month follow-up assessment
  Question asks: How long do you typically wait to drive after using alcohol and Cannabis used at the same time so that the effects overlap. Participants answer in hours and minutes which is transformed into total number of minutes.
Reported wait time to drive after using alcohol measured in minutes at 6 month follow up | From 3 months after baseline to 3 months later at 6 month follow-up assessment
  Question asks: How long do you typically wait to drive after using alcohol . Participants answer in hours and minutes which is transformed into total number of minutes.
Reported wait time to drive after using cannabis measured in minutes at 6 month follow up | From 3 months after baseline to 3 months later at 6 month follow-up assessment
  Question asks: How long do you typically wait to drive after using cannabis. Participants answer in hours and minutes which is transformed into total number of minutes.

IPD SHARING:
Plan to Share IPD: Undecided